CLINICAL TRIAL: NCT00444600
Title: Intravitreal Ranibizumab or Triamcinolone Acetonide in Combination With Laser Photocoagulation for Diabetic Macular Edema
Brief Title: Laser-Ranibizumab-Triamcinolone for Diabetic Macular Edema
Acronym: LRT for DME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Allergan (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-133; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Diabetic Retinopathy; Diabetic Macular Edema; Lucentis; Ranibizumab; Triamcinolone; Laser photocoagulation; Combination Therapy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Triamcinolone Acetonide; Lasers; Adrenal Cortex Hormones; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.5mg Ranibizumab plus laser (Experimental)
  Interventions: Drug: Ranibizumab + laser
- 0.5 mg Ranibizumab plus deferred laser (Experimental)
  Interventions: Drug: Ranibizumab + deferred laser
- 4 mg Triamcinolone plus laser (Experimental)
  Interventions: Drug: Triamcinolone Acetonide + laser
- Sham plus laser (Active Comparator)
  Interventions: Drug: Sham injection + laser

INTERVENTIONS:
Drug: Triamcinolone Acetonide + laser — 4 mg intravitreal triamcinolone at randomization plus focal photocoagulation 1 week post-injection, repeated every 16 weeks with sham injections at 4-week intervals in-between. Retreatment starting at 16 weeks depends on visual acuity and OCT.
  Other Names: corticosteroid
  Arms: 4 mg Triamcinolone plus laser
Drug: Ranibizumab + laser — 0.5 mg intravitreal ranibizumab at randomization plus focal photocoagulation 1 week post-injection. Injections are repeated every 4 weeks with focal photocoagulation given post-injection every 16 weeks. Retreatment starting at 16 weeks depends on visual acuity and OCT.
  Other Names: Lucentis, anti-VEGF drug
  Arms: 0.5mg Ranibizumab plus laser
Drug: Sham injection + laser — Sham injection at randomization plus focal photocoagulation 1 week post-injection. Injections are repeated every 4 weeks with focal photocoagulation given post-injection every 16 weeks. Retreatment starting at 16 weeks depends on visual acuity and OCT.
  Other Names: placebo
  Arms: Sham plus laser
Drug: Ranibizumab + deferred laser — 0.5 mg intravitreal ranibizumab at randomization, repeated every 4 weeks. Retreatment starting at 16 weeks depends on visual acuity and OCT. If improvement has not occured from injections alone, laser can be given starting at the 24 week visit.
  Other Names: Lucentis, anti-VEGF drug
  Arms: 0.5 mg Ranibizumab plus deferred laser

SUMMARY:
The purpose of the study is to find out which is a better treatment for diabetic macular edema (DME): laser alone, laser combined with an intravitreal injection of triamcinolone, laser combined with an intravitreal injection of ranibizumab, or intravitreal injection of ranibizumab alone. At the present time, it is not known whether intravitreal steroid or anti-vascular endothelial growth factor (anti-VEGF) injections, with or without laser treatment, are better than just laser by itself. It is possible that one or both of the types of injections, with or without laser treatment, will improve vision more often than will laser without injections. However, even if better vision outcomes are seen with injections, side effects may be more of a problem with the injections than with laser. Therefore, this study is conducted to find out whether the benefits of the injections will outweigh the risks.

DETAILED DESCRIPTION:
Thus far the only demonstrated means to reduce the risk of vision loss from diabetic macular edema are laser photocoagulation, intensive glycemic control, and blood pressure control. Earlier studies have shown that photocoagulation, although effective in reducing the risk of moderate vision loss, can eventually result in retinal and retinal pigment epithelium atrophy resulting in loss of central vision, central scotomata, and decreased color vision. Consequently, many retinal specialists today tend to treat diabetic macular edema (DME) with lighter, less intense laser burns than was originally specified in the Early Treatment Diabetic Retinopathy Study (ETDRS). The additional unsatisfactory outcome from treatments with laser photocoagulation in a significant proportion of eyes with DME has prompted interest in other treatment modalities. One such treatment is pars plana vitrectomy. Studies suggest that vitreomacular traction may play a role in increased retinal vascular permeability, and that removal of the vitreous, or relief of mechanical traction with vitrectomy and membrane stripping may substantially improve macular edema and visual acuity. However, this treatment may be applicable only to a specific subset of eyes with a component of vitreomacular traction secondary to edema. Other treatment modalities such as pharmacologic therapy with oral protein kinase C inhibitors and intravitreal corticosteroids are under investigation.

The use of antibodies targeted at vascular endothelial growth factor (VEGF) is another treatment modality that needs to be further explored for its potential benefits. Increased VEGF levels have been demonstrated in the retina and vitreous of human eyes with diabetic retinopathy. VEGF, also knows as vascular permeability factor, has been shown to increase retinal vascular permeability in in vivo models. Therapy that inhibits VEGF, therefore, may represent a useful therapeutic modality which targets the underlying pathogenesis of diabetic macular edema. Ranibizumab is a promising anti-VEGF drug. Its efficacy and safety have been demonstrated in treatment of age-related macular degeneration. Reports of its use and that of other anti-VEGF drugs in DME have suggested sufficient benefit to warrant evaluation of efficacy and safety in a phase III trial. Corticosteroids, a class of substances with anti-inflammatory properties, have also been demonstrated to inhibit the expression of the VEGF gene. The Diabetic Retinopathy Clinical Research Network (DRCR.net) is currently conducting a phase III randomized clinical trial comparing focal photocoagulation to intravitreal corticosteroids (triamcinolone acetonide) for diabetic macular edema. However, even if triamcinolone or ranibizumab are proven to be efficacious, a major concern, based on clinical observations with intravitreal corticosteroids, is that DME will recur as the effect of the intravitreal drug wears off, necessitating repetitive injections long-term. Combining an intravitreal drug (triamcinolone or ranibizumab) with photocoagulation provides hope that one could get the short-term benefit of the intravitreal drug (decreased retinal thickening and decreased fluid leakage) and the long-term reduction in fluid leakage as a result of photocoagulation. In addition, it is possible that the worsening of macular edema immediately following focal photocoagulation, a known complication of this treatment, could be decreased if an intravitreal drug was present at the time of photocoagulation. This might result in an increased likelihood of vision improvement following photocoagulation and a decreased likelihood of vision loss.

This study is designed to determine if ranibizumab alone or ranibizumab added to laser photocoagulation is more efficacious than photocoagulation alone, and if so, to determine if combining ranibizumab with photocoagulation reduces the total number of injections needed to obtain these benefits. Furthermore, this study is designed to determine if combining photocoagulation with corticosteroids, the only other class of drugs currently being considered for treatment of DME, is efficacious in the population being enrolled.

Subjects will be randomly assigned to one of the following 4 groups:

1. Group A: Sham injection plus focal (macular) photocoagulation
2. Group B: 0.5 mg injection of intravitreal ranibizumab plus focal photocoagulation
3. Group C: 0.5 mg injection of intravitreal ranibizumab plus deferred focal photocoagulation
4. Group D: 4 mg intravitreal triamcinolone plus focal photocoagulation

In groups A, B and D, laser will be given 7-10 days after the initial injection at the time of the injection follow-up safety visit. During the first year, subjects are evaluated for retreatment every 4 weeks. The injection for group A is a sham and for groups B and C ranibizumab. For group D, a triamcinolone injection is given if one has not been given in the prior 15 weeks; otherwise a sham injection is given. For Groups A, B, and D, focal photocoagulation will be given 7 to 10 days later following each injection unless focal photocoagulation has been given in the past 15 weeks or no macular edema is present. In Years 2 and 3, subjects continue to be evaluated for retreatment every 4 weeks unless injections are discontinued due to failure. In that case, follow-up visits occur every 4 months and treatment is at investigator discretion.

ELIGIBILITY:
General Inclusion Criteria

To be eligible, the following inclusion criteria (1-5) must be met:

* Age >= 18 years
* Diagnosis of diabetes mellitus (type 1 or type 2)
* At least one eye meets the study eye criteria
* Fellow eye (if not a study eye) meets criteria
* Able and willing to provide informed consent

General Exclusion Criteria

A subject is not eligible if any of the following exclusion criteria are present:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry.
* Known allergy to any component of the study drug.
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
* Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.
* Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
* Systemic anti-vascular growth factor (anti-VEGF) or pro-VEGF treatment within 4 months prior to randomization.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months.
* Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the first 12 months of the study.

Study Eye Inclusion Criteria

The subject must have one eye meeting all of the inclusion criteria and none of the exclusion criteria listed below. A subject may have two study eyes only if both are eligible at the time of randomization.

* Best corrected electronic Early Treatment Diabetic Retinopathy (E-ETDRS) visual acuity letter score <= 78 (i.e., 20/32 or worse) and >= 24 (i.e., 20/320 or better) within 8 days of randomization.
* On clinical exam, definite retinal thickening due to diabetic macular edema involving the center of the macula.
* Ocular coherence tomography (OCT) central subfield >=250 microns within 8 days of randomization.
* Media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs.
* If prior macular photocoagulation has been performed, the investigator believes that the study eye may possibly benefit from additional photocoagulation.

Study Eye Exclusion Criteria

The following exclusions apply to the study eye only (i.e., they may be present for the nonstudy eye):

* Macular edema is considered to be due to a cause other than diabetic macular edema.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition).
* An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.)
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of treatment for diabetic macular edema at any time in the past 4 months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, anti-VEGF drugs, or any other treatment).
* History of panretinal (scatter) photocoagulation (PRP) within 4 months prior to randomization.
* Anticipated need for PRP in the 6 months following randomization.
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
* History of yttrium aluminum garnet (YAG) capsulotomy performed within 2 months prior to randomization.
* Aphakia.
* Intraocular pressure >= 25 mmHg.
* History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: history of angle-closure glaucoma is not an exclusion criterion).
* History of steroid-induced intraocular pressure (IOP) elevation that required IOP-lowering treatment.
* History of prior herpetic ocular infection.
* Exam evidence of ocular toxoplasmosis.
* Exam evidence of pseudoexfoliation.
* Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 691 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Elman, M.D., Study Chair — Elman Retina Group, PA
Locations (50):
- United States (50):
  - Sall Research Medical Center, Artesia, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of California, Irvine, Irvine, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Vitreous Consultants, Fort Lauderdale, Florida
  - Retina Consultants of Southwest Florida, Fort Myers, Florida
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Illinois Retina Associates, Joliet, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Medical Associates Clinic, P.C., Dubuque, Iowa
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Retina Consultants of Delmarva, P.A., Salisbury, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Retina Center, PA, Minneapolis, Minnesota
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - University of North Carolina, Dept of Ophthalmology, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Retina Consultants, Providence, Rhode Island
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - West Texas Retina Consultants P.A., Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Elman MJ, Bressler NM, Qin H, Beck RW, Ferris FL 3rd, Friedman SM, Glassman AR, Scott IU, Stockdale CR, Sun JK; Diabetic Retinopathy Clinical Research Network. Expanded 2-year follow-up of ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):609-14. doi: 10.1016/j.ophtha.2010.12.033. PMID 21459214
- [Background] Diabetic Retinopathy Clinical Research Network; Writing Committee; Aiello LP, Beck RW, Bressler NM, Browning DJ, Chalam KV, Davis M, Ferris FL 3rd, Glassman AR, Maturi RK, Stockdale CR, Topping TM. Rationale for the diabetic retinopathy clinical research network treatment protocol for center-involved diabetic macular edema. Ophthalmology. 2011 Dec;118(12):e5-14. doi: 10.1016/j.ophtha.2011.09.058. PMID 22136692
- [Background] Glassman AR, Stockdale CR, Beck RW, Baker C, Bressler NM; Diabetic Retinopathy Clinical Research Network. Evaluation of masking study participants to intravitreal injections in a randomized clinical trial. Arch Ophthalmol. 2012 Feb;130(2):190-4. doi: 10.1001/archophthalmol.2011.387. PMID 22332211
- [Background] Bressler SB, Qin H, Beck RW, Chalam KV, Kim JE, Melia M, Wells JA 3rd; Diabetic Retinopathy Clinical Research Network. Factors associated with changes in visual acuity and central subfield thickness at 1 year after treatment for diabetic macular edema with ranibizumab. Arch Ophthalmol. 2012 Sep;130(9):1153-61. doi: 10.1001/archophthalmol.2012.1107. PMID 22965591
- [Background] Bressler SB, Qin H, Melia M, Bressler NM, Beck RW, Chan CK, Grover S, Miller DG; Diabetic Retinopathy Clinical Research Network. Exploratory analysis of the effect of intravitreal ranibizumab or triamcinolone on worsening of diabetic retinopathy in a randomized clinical trial. JAMA Ophthalmol. 2013 Aug;131(8):1033-40. doi: 10.1001/jamaophthalmol.2013.4154. PMID 23807371
- [Background] Bressler SB, Almukhtar T, Aiello LP, Bressler NM, Ferris FL 3rd, Glassman AR, Greven CM; Diabetic Retinopathy Clinical Research Network. Green or yellow laser treatment for diabetic macular edema: exploratory assessment within the Diabetic Retinopathy Clinical Research Network. Retina. 2013 Nov-Dec;33(10):2080-8. doi: 10.1097/IAE.0b013e318295f744. PMID 23792486
- [Background] Bressler SB, Almukhtar T, Bhorade A, Bressler NM, Glassman AR, Huang SS, Jampol LM, Kim JE, Melia M; Diabetic Retinopathy Clinical Research Network Investigators. Repeated intravitreous ranibizumab injections for diabetic macular edema and the risk of sustained elevation of intraocular pressure or the need for ocular hypotensive treatment. JAMA Ophthalmol. 2015 May;133(5):589-97. doi: 10.1001/jamaophthalmol.2015.186. PMID 25719991
- [Background] Bressler SB, Odia I, Glassman AR, Danis RP, Grover S, Hampton GR, Jampol LM, Maguire MG, Melia M. CHANGES IN DIABETIC RETINOPATHY SEVERITY WHEN TREATING DIABETIC MACULAR EDEMA WITH RANIBIZUMAB: DRCR.net Protocol I 5-Year Report. Retina. 2018 Oct;38(10):1896-1904. doi: 10.1097/IAE.0000000000002302. PMID 30234859
- [Background] Bressler SB, Melia M, Glassman AR, Almukhtar T, Jampol LM, Shami M, Berger BB, Bressler NM; Diabetic Retinopathy Clinical Research Network. RANIBIZUMAB PLUS PROMPT OR DEFERRED LASER FOR DIABETIC MACULAR EDEMA IN EYES WITH VITRECTOMY BEFORE ANTI-VASCULAR ENDOTHELIAL GROWTH FACTOR THERAPY. Retina. 2015 Dec;35(12):2516-28. doi: 10.1097/IAE.0000000000000617. PMID 26035510
- [Background] Bressler SB, Ayala AR, Bressler NM, Melia M, Qin H, Ferris FL 3rd, Flaxel CJ, Friedman SM, Glassman AR, Jampol LM, Rauser ME; Diabetic Retinopathy Clinical Research Network. Persistent Macular Thickening After Ranibizumab Treatment for Diabetic Macular Edema With Vision Impairment. JAMA Ophthalmol. 2016 Mar;134(3):278-85. doi: 10.1001/jamaophthalmol.2015.5346. PMID 26746868
- [Result] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Result] Diabetic Retinopathy Clinical Research Network; Elman MJ, Qin H, Aiello LP, Beck RW, Bressler NM, Ferris FL 3rd, Glassman AR, Maturi RK, Melia M. Intravitreal ranibizumab for diabetic macular edema with prompt versus deferred laser treatment: three-year randomized trial results. Ophthalmology. 2012 Nov;119(11):2312-8. doi: 10.1016/j.ophtha.2012.08.022. Epub 2012 Sep 19. PMID 22999634
- [Result] Bressler SB, Glassman AR, Almukhtar T, Bressler NM, Ferris FL, Googe JM Jr, Gupta SK, Jampol LM, Melia M, Wells JA 3rd; Diabetic Retinopathy Clinical Research Network. Five-Year Outcomes of Ranibizumab With Prompt or Deferred Laser Versus Laser or Triamcinolone Plus Deferred Ranibizumab for Diabetic Macular Edema. Am J Ophthalmol. 2016 Apr;164:57-68. doi: 10.1016/j.ajo.2015.12.025. Epub 2016 Jan 21. PMID 26802783
- [Result] Elman MJ, Ayala A, Bressler NM, Browning D, Flaxel CJ, Glassman AR, Jampol LM, Stone TW; Diabetic Retinopathy Clinical Research Network. Intravitreal Ranibizumab for diabetic macular edema with prompt versus deferred laser treatment: 5-year randomized trial results. Ophthalmology. 2015 Feb;122(2):375-81. doi: 10.1016/j.ophtha.2014.08.047. Epub 2014 Oct 28. PMID 25439614
- [Derived] Talcott KE, Valentim CCS, Hill L, Stoilov I, Singh RP. Baseline Diabetic Retinopathy Severity and Time to Diabetic Macular Edema Resolution with Ranibizumab Treatment: A Meta-Analysis. Ophthalmol Retina. 2023 Jul;7(7):605-611. doi: 10.1016/j.oret.2023.02.003. Epub 2023 Feb 10. PMID 36774994
- [Derived] Gangaputra S, Almukhtar T, Glassman AR, Aiello LP, Bressler N, Bressler SB, Danis RP, Davis MD; Diabetic Retinopathy Clinical Research Network. Comparison of film and digital fundus photographs in eyes of individuals with diabetes mellitus. Invest Ophthalmol Vis Sci. 2011 Aug 3;52(9):6168-73. doi: 10.1167/iovs.11-7321. PMID 21571677
- [Derived] Bhavsar AR, Googe JM Jr, Stockdale CR, Bressler NM, Brucker AJ, Elman MJ, Glassman AR; Diabetic Retinopathy Clinical Research Network. Risk of endophthalmitis after intravitreal drug injection when topical antibiotics are not required: the diabetic retinopathy clinical research network laser-ranibizumab-triamcinolone clinical trials. Arch Ophthalmol. 2009 Dec;127(12):1581-3. doi: 10.1001/archophthalmol.2009.304. PMID 20008710
- See also: DRCR Retina Network — https://public.jaeb.org/drcrnet/pubs

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty two academic and community based sites across the United States recruited 691 study participants from March 2007 to December 2008.
Pre-assignment Details: Participants with two study eyes enrolled each eye in a different treatment group. Therefore, each treatment group/arm includes no more than one study eye for a given participant, and thus the numbers of eyes is equal to the number of participants in each arm.
Groups:
- Sham+Prompt Laser: Sham injection at randomization plus focal photocoagulation 1 week post-injection. Injections are repeated every 4 weeks with focal photocoagulation given post-injection every 16 weeks. Retreatment starting at 16 weeks depends on visual acuity and OCT.
- 0.5 mg Ranibizumab+Prompt Laser: 0.5 mg intravitreal ranibizumab at randomization plus focal photocoagulation 1 week post-injection. Injections are repeated every 4 weeks with focal photocoagulation given post-injection every 16 weeks. Retreatment starting at 16 weeks depends on visual acuity and OCT.
- 0.5 mg Ranibizumab+Deferred Laser: 0.5 mg intravitreal ranibizumab at randomization, repeated every 4 weeks. Retreatment starting at 16 weeks depends on visual acuity and OCT. If improvement has not occured from injections alone, laser can be given starting at the 24 week visit.
- 4 mg Triamcinolone+Prompt Laser: 4 mg intravitreal triamcinolone at randomization plus focal photocoagulation 1 week post-injection, repeated every 16 weeks with sham injections at 4-week intervals in-between. Retreatment starting at 16 weeks depends on visual acuity and OCT.
Period: Overall Study
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Started | 293 (Number of eyes) | 187 (Number of eyes) | 188 (Number of eyes) | 186 (Number of eyes)
Completed | 274 (Number of eyes) | 171 (Number of eyes) | 178 (Number of eyes) | 176 (Number of eyes)
Not Completed | 19 | 16 | 10 | 10
Not completed — Death | 7 | 5 | 3 | 2
Not completed — Dropped | 11 | 11 | 7 | 7
Not completed — Missed visit | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser | Total
Number analyzed (Participants) | 293 | 187 | 188 | 186 | 854
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [57 to 69] | 62 [56 to 70] | 64 [58 to 70] | 62 [55 to 70] | 63 [56 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 85 | 78 | 86 | 372
  Male | 170 | 102 | 110 | 100 | 482
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 202 | 131 | 134 | 134 | 601
  African American | 51 | 30 | 25 | 32 | 138
  Hispanic or Latino | 34 | 21 | 25 | 15 | 95
  Asian | 4 | 1 | 2 | 4 | 11
  Native Hawaiian/Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  More than one race | 1 | 1 | 1 | 0 | 3
  Unknown/not reported | 1 | 2 | 1 | 1 | 5
Visual Acuity Letter Score (approximate Snellen equivalent) by randomization strata [Number; unit: Eyes]
  ≥66 (better than 20/50) | 146 | 95 | 95 | 93 | 429
  ≤65 (20/50 or worse) | 147 | 92 | 93 | 93 | 425
Classification of diabetic macular edema [Number; unit: Eyes] — Based on clinical exam.
  Eyes
    Predominantly focal | 78 | 60 | 68 | 53 | 259
    Neither predominantly focal or diffuse | 71 | 46 | 41 | 48 | 206
    Predominantly diffuse | 144 | 81 | 79 | 85 | 389
Number of study eyes [Number; unit: Participants]
  1 study eye | 130 | 131 | 132 | 135 | 528
  2 study eyes | 163 | 56 | 56 | 51 | 326
Diabetes Type [Number; unit: Participants]
  Type 1 | 25 | 11 | 15 | 14 | 65
  Type 2 | 260 | 172 | 170 | 166 | 768
  Uncertain | 8 | 4 | 3 | 6 | 21
Duration of diabetes [Median (Inter-Quartile Range); unit: Years] | 16 [9 to 22] | 18 [12 to 24] | 17 [11 to 22] | 17 [11 to 24] | 16 [10 to 23]
HbA1c [Median (Inter-Quartile Range); unit: Percentage] — Missing HbA1c data for 17, 3, 7 and 8 study participants in the sham+prompt laser, ranibizumab+prompt laser, ranibizumab+deferred laser and triamcinolone+prompt laser groups, respectively.
  Percentage | 7.3 [6.6 to 8.3] | 7.3 [6.6 to 8.4] | 7.5 [6.7 to 8.4] | 7.4 [6.5 to 8.6] | 7.3 [6.6 to 8.4]
Prior cardiovascular event [Number; unit: Participants] — Based on medical history of condition.
  Participants
    Yes | 93 | 66 | 61 | 61 | 281
    No | 200 | 121 | 127 | 125 | 573
Hypertension [Number; unit: Participants]
  Yes | 240 | 154 | 156 | 148 | 698
  No | 53 | 33 | 32 | 38 | 156
Prior Panretinal Photocoagulation [Number; unit: Eyes]
  Yes | 48 | 36 | 31 | 37 | 152
  No | 245 | 151 | 157 | 149 | 702
Prior treatment for diabetic macular edema [Number; unit: Eyes]
  No | 105 | 74 | 74 | 61 | 314
  Yes | 188 | 113 | 114 | 125 | 540
Prior laser for diabetic macular edema [Number; unit: Eyes]
  Yes | 173 | 101 | 101 | 114 | 489
  No | 120 | 86 | 87 | 72 | 365
Prior IVT for diabetic macular edema [Number; unit: Eyes] — IVT = intravitreal triamcinolone
  Eyes
    Yes | 39 | 22 | 36 | 31 | 128
    No | 254 | 165 | 152 | 155 | 726
Prior vitrectomy for diabetic macular edema [Number; unit: Eyes]
  Yes | 15 | 7 | 5 | 12 | 39
  No | 278 | 180 | 183 | 174 | 815
Prior peribulbar triamcinolone for diabetic macular edema [Number; unit: Eyes]
  Yes | 12 | 9 | 5 | 5 | 31
  No | 281 | 178 | 183 | 181 | 823
Prior anti-VEGF for diabetic macular edema [Number; unit: Eyes] — VEGF = vascular endothelial growth factor
  Eyes
    Yes | 24 | 24 | 21 | 20 | 89
    No | 269 | 163 | 167 | 166 | 765
Intraocular pressure [Median (Inter-Quartile Range); unit: mmHg] | 16 [14 to 18] | 16 [14 to 18] | 16 [14 to 18] | 16 [14 to 18] | 16 [14 to 18]
Currently on intraocular pressure lowering medicine for glaucoma or ocular hypertension [Number; unit: Eyes]
  Yes | 5 | 6 | 4 | 2 | 17
  No | 288 | 181 | 184 | 184 | 837
Lens status [Number; unit: Eyes] — Based on clinical exam.
  Eyes
    Phakic | 192 | 131 | 134 | 124 | 581
    Anterior Chamber Intraocular Lense | 3 | 1 | 1 | 0 | 5
    Posterior Chamber Intraocular Lense | 98 | 55 | 53 | 62 | 268
E-ETDRS Visual Acuity Letter Score [Median (Inter-Quartile Range); unit: Letter Score] — Best corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. Best value on the scale 97, worst 0.
  Letter Score | 65 [56 to 73] | 66 [55 to 72] | 66 [58 to 72] | 66 [57 to 72] | 66 [56 to 72]
Central subfield thickness on optical coherence tomography [Median (Inter-Quartile Range); unit: microns] | 407 [309 to 505] | 371 [302 to 464] | 382 [298 to 488] | 374 [298 to 463] | 381 [306 to 485]
Retinal volume on optical coherence tomography [Median (Inter-Quartile Range); unit: microns] | 8.7 [7.8 to 10.0] | 8.4 [7.5 to 9.6] | 8.4 [7.4 to 9.8] | 8.5 [7.8 to 9.7] | 8.5 [7.7 to 9.7]
Optical coherence tomography cystoid abnormality [Number; unit: Eyes]
  No evidence | 19 | 13 | 12 | 8 | 52
  Questionable or definite | 274 | 171 | 174 | 177 | 796
  Cannot grade or missing | 0 | 3 | 2 | 1 | 6
Optical coherence tomography subretinal fluid present [Number; unit: Eyes]
  No evidence | 222 | 149 | 140 | 146 | 657
  Questionable or definite | 70 | 36 | 45 | 38 | 189
  Cannot grade | 1 | 2 | 3 | 2 | 8
ETDRS retinopathy severity level (ETDRS description) [Number; unit: Eyes] — ETDRS = Early Treatment Diabetic Retinopathy Study; DR = diabetic retinopathy; PDR = proliferative diabetic retinopathy.
  Criteria are based on the ETDRS fundus photographic risk factors for the progression of diabetic retinopathy. ETDRS report no. 12. Ophthalmology 1991; 98:823-833
  Eyes
    Diabetic retinopathy absent | 5 | 4 | 3 | 1 | 13
    Minimal non-proliferative DR | 2 | 2 | 3 | 3 | 10
    Mild to moderately severe non-proliferative DR | 171 | 103 | 107 | 95 | 476
    Severe non-proliferative DR | 22 | 16 | 11 | 15 | 64
    Scars of full or partial PRP present;PDR absent | 38 | 30 | 30 | 29 | 127
    Mild to moderate proliferative DR | 33 | 24 | 22 | 34 | 113
    High risk proliferative DR | 7 | 4 | 1 | 3 | 15
    Cannot grade | 10 | 1 | 2 | 4 | 17
    Missing | 5 | 3 | 9 | 2 | 19

OUTCOME MEASURES:

1. Secondary Outcome: Change in Retinal Thickening of Central Subfield on Optical Coherence Tomography From Baseline to 1 Year
Description: Negative change denotes an improvement.
Time Frame: from baseline to 1 year
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 271 | 171 | 175 | 173
Number analyzed (Eyes) | 271 | 171 | 175 | 173
microns | -102 (151) | -131 (129) | -137 (136) | -127 (140)
Statistical Analysis 1: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Difference in central subfield thickness mean change from sham+prompt laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Confidence intervals are adjusted for multiple comparisons; Adjusted for baseline retinal thickness and visual acuity and correlation between two study eyes; Difference in mean change = -55, 95% CI 2-sided [-78 to -32]
Statistical Analysis 2: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Difference in optical coherence tomography central subfield thickness mean change from sham+prompt laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Confidence intervals are adjusted for multiple comparisons; Adjusted for baseline retinal thickness and visual acuity and correlation between two study eyes; Difference in mean change = -49, 95% CI 2-sided [-72 to -26]
Statistical Analysis 3: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Difference in optical coherence tomography central subfield thickness mean change from sham+prompt laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Confidence interval is adjusted for multiple comparisons; Adjusted for baseline retinal thickness and visual acuity and correlation between two study eyes; Difference in mean change = -52, 95% CI 2-sided [-75 to -29]

2. Secondary Outcome: Number of Injections in First Year
Description: Maximum possible number of injections for each of the following groups: sham+prompt laser=13 sham injections;ranibizumab+prompt laser=13 ranibizumab injections; ranibizumab+deferred laser=13 ranibizumab injections; triamcinolone+prompt laser=4 triamcinolone injections and 9 sham injections.
Time Frame: from baseline to 1 year
Population: Sham+prompt laser group listed median excludes 56 eyes among 163 participants with 2 study eyes that were unmasked at baseline because the participant's other eye was in the ranibizumab+deferred laser group, precluding sham injections for the study eye assigned to sham+prompt laser.
Measure: Median (Inter-Quartile Range); unit: Injections
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 274 | 171 | 178 | 176
Number analyzed (Eyes) | 274 | 171 | 178 | 176
Injections | 11 [8 to 13] | 8 [6 to 10] | 9 [6 to 11] | 3 [2 to 4]

3. Primary Outcome: Mean Change in Visual Acuity (Letters) From Baseline to 1 Year Adjusted for Baseline Visual Acuity
Description: Change in best correct visual acuity letter score from baseline to one year as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. A positive change denotes an improvement. Best value on the scale 97, worst 0.
Time Frame: from baseline to 1 Year
Population: For eyes without any 1-year data the last observation carried forward method was used to impute data for the primary analysis. followed intention to treat principle.
Measure: Mean (Standard Deviation); unit: Letters
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
Letters | 3 (13) | 9 (11) | 9 (12) | 4 (13)
Statistical Analysis 1: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted for multiple comparisons; Adjusted for baseline visual acuity and correlation between 2 study eyes; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [3.2 to 8.5]
Statistical Analysis 2: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted for multiple comparisons; Adjusted for baseline visual acuity and correlation between 2 study eyes; Mean Difference (Final Values) = 6.0, 95% CI 2-sided [3.4 to 8.6]
Statistical Analysis 3: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Test type: Superiority or Other; p = 0.31, ANCOVA — Adjusted for multiple comparisons; Adjusted for baseline visual acuity and correlation between 2 study eyes; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-1.5 to 3.7]

4. Primary Outcome: Distribution of Change in Visual Acuity (Letters) From Baseline to 1 Year
Description: Change in best correct visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method.
Time Frame: from baseline to 1 Year
Population: For eyes without any 1-year data the last observation carried forward method was used to impute data for the primary analysis.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
Eyes
  ≥15 letter improvement | 43 | 57 | 52 | 39
  14-10 letter improvement | 38 | 38 | 36 | 22
  9-5 letter improvement | 67 | 34 | 54 | 32
  Same ±4 letters | 86 | 38 | 35 | 54
  5-9 letters worse | 20 | 14 | 5 | 12
  10-14 letters worse | 16 | 3 | 2 | 12
  ≥15 letters worse | 23 | 3 | 4 | 15
Statistical Analysis 1: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Difference in proportion with ≥10 letter improvement for sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = 23, 95% CI 2-sided [13 to 34]
Statistical Analysis 2: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Difference in proportion with ≥10 letter improvement from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial regression — Confidence intervals adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = 19, 95% CI 2-sided [9 to 29]
Statistical Analysis 3: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Difference in proportion with ≥10 letter improvement from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial regression — Confidence intervals adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = 6, 95% CI 2-sided [-4 to 16]
Statistical Analysis 4: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Relative risk for ≥10 letter improvement comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p < 0.001, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.84, 95% CI 2-sided [1.40 to 2.42]
Statistical Analysis 5: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Relative risk for ≥10 letter improvement comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p < 0.001, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.68, 95% CI 2-sided [1.27 to 2.21]
Statistical Analysis 6: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Relative risk for ≥10 letter improvement comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p = 0.16, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.88 to 1.66] — Eyes were analyzed
Statistical Analysis 7: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Difference in proportion with ≥10 letter worsening from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = -10, 95% CI 2-sided [-16 to -5]
Statistical Analysis 8: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Difference in proportion with ≥10 letter worsening from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = -10, 95% CI 2-sided [-16 to -4]
Statistical Analysis 9: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Difference in proportion with ≥10 letter worsening from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = 1, 95% CI 2-sided [-7 to 9]
Statistical Analysis 10: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Relative risk for ≥10 letter worsening comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p < 0.001, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 0.24, 95% CI 2-sided [0.09 to 0.65]
Statistical Analysis 11: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Relative risk for ≥10 letter worsening comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p = 0.001, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 0.24, 95% CI 2-sided [0.08 to 0.68]
Statistical Analysis 12: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Relative risk for ≥10 letter worsening comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p = 0.75, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.62 to 1.87]
Statistical Analysis 13: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Difference in proportion with ≥15 letter improvement from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between to study eyes; Proportion = 16, 95% CI 2-sided [6 to 26]
Statistical Analysis 14: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Difference in proportion with ≥15 letter improvement from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = 13, 95% CI 2-sided [4 to 22]
Statistical Analysis 15: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Difference in proportion with ≥15 letter improvement from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = 6, 95% CI 2-sided [-2 to 15]
Statistical Analysis 16: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Relative risk for ≥15 letter improvement comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p < 0.001, Log-Binomial Regression; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 2.09, 95% CI 2-sided [1.35 to 3.22]
Statistical Analysis 17: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Relative risk for ≥15 letter improvement comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p < 0.001, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.89, 95% CI 2-sided [1.25 to 2.87]
Statistical Analysis 18: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Relative risk for ≥15 letter improvement comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p = 0.07, Log-Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.43, 95% CI 2-sided [0.90 to 2.29]
Statistical Analysis 19: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Difference in proportion with ≥15 letter worsening from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = -6, 95% CI 2-sided [-11 to -2]
Statistical Analysis 20: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Difference in proportion with ≥15 letter worsening from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = -6, 95% CI 2-sided [-10 to -1]
Statistical Analysis 21: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Difference in proportion with ≥15 letter worsening from sham+prompt laser at 1 year; Test type: Superiority or Other; Binomial Regression — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Proportion = 0, 95% CI 2-sided [-6 to 6]
Statistical Analysis 22: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Relative risk for ≥15 letter worsening comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p = 0.009, Log-Binomial Regression; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 0.21, 95% CI 2-sided [0.05 to 0.87]
Statistical Analysis 23: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Relative risk for ≥15 letter worsening comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p = 0.01, Log-Binomial Regression; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 0.28, 95% CI 2-sided [0.08 to 0.97]
Statistical Analysis 24: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Relative risk for ≥15 letter worsening comparison with sham+prompt laser at 1 year; Test type: Superiority or Other; p = 0.95, Log-Binomial Regression; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.47 to 2.20]

5. Other Pre Specified Outcome: Central Subfield Thickness < 250 With at Least a 25 Micron Decrease From Baseline to 1 Year
Time Frame: 1 Year
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 271 | 171 | 175 | 173
Number analyzed (Eyes) | 271 | 171 | 175 | 173
Eyes | 72 | 91 | 74 | 82
Statistical Analysis 1: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Relative risk for comparison with sham+prompt laser; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Confidence intervals are adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 2.00, 95% CI 2-sided [1.52 to 2.64]
Statistical Analysis 2: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Relative risk for comparison with sham+prompt laser; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Confidence intervals adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.55, 95% CI 2-sided [1.13 to 2.13]
Statistical Analysis 3: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Relative risk for comparison with sham+prompt laser; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Confidence intervals adjusted for multiple comparisons; Adjusted for correlation between 2 study eyes and multiple comparisons; Risk Ratio (RR) = 1.76, 95% CI [1.31 to 2.36]

6. Other Pre Specified Outcome: Distribution of Logarithmic Transformation of Optical Coherence Tomography (LogOCT) Improvement and Worsening
Description: Logarithmic transformation of optical coherence tomography central subfield thickness is calculated by taking the log base 10 of the ratio of the central subfield thickness divided by 200 and rounding to the nearest hundredth. The change is the change in the log values.
Time Frame: 1 Year
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 271 | 171 | 175 | 173
Number analyzed (Eyes) | 271 | 171 | 175 | 173
Eyes
  ≥2 step improvement | 81 | 72 | 71 | 65
  ≥2 step worsening | 6 | 1 | 0 | 4

7. Primary Outcome: Change in Visual Acuity From Baseline to 1 Year Among Eyes That Were Pseudophakic at Baseline
Time Frame: from baseline to 1 Year
Measure: Mean (Standard Deviation); unit: Letters
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
Letters
  Not pseudophakic at baseline | 2 (13) | 9 (10) | 10 (14) | 2 (14)
  Pseudophakic at baseline | 4 (14) | 8 (12) | 7 (9) | 8 (9)

8. Primary Outcome: Change in Visual Acuity From Baseline to 1 Year Among Eyes That Had Prior Treatment for Diabetic Macular Edema
Time Frame: from baseline to 1 Year
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Letters
  No | 2 (14) | 9 (12) | 11 (13) | 3 (13)
  Yes | 3 (13) | 9 (10) | 8 (12) | 5 (13)

9. Primary Outcome: Change in Visual Acuity From Baseline to 1 Year Grouped by Baseline Visual Acuity Letter Score
Description: Change in best correct visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the Early Treatment Diabetic Retinopathy Study (ETDRS) method. A positive change denotes an improvement. Best value on the scale 97, worst 0.
Time Frame: from baseline to 1 Year
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Letters
  ≥66 (better than 20/50) | 1 (12) | 6 (10) | 5 (13) | 1 (11)
  ≤65 (20/50 or worse) | 5 (14) | 12 (11) | 13 (10) | 7 (14)

10. Primary Outcome: Change in Visual Acuity From Baseline to 1 Year Grouped by Optical Coherence Tomography Central Subfield Thickness
Description: as for outcome 3
Time Frame: from baseline to 1 Year
Measure: Mean (Standard Deviation); unit: Letters
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
Letters
  <400 microns | 3 (11) | 7 (11) | 7 (12) | 3 (12)
  ≥400 microns | 3 (15) | 11 (10) | 11 (13) | 6 (14)

11. Primary Outcome: Change in Visual Acuity From Baseline to 1 Year Grouped by Diabetic Retinopathy Severity
Description: as for outcome 3
Time Frame: from baseline to 1 Year
Measure: Mean (Standard Deviation); unit: Letters
Units Other Than Participants: eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (eyes) | 293 | 187 | 188 | 186
Letters
  Moderately severe non-proliferative DR or better | 3 (13) | 10 (11) | 9 (12) | 3 (14)
  Severe non-proliferative DR or worse | 2 (15) | 8 (10) | 9 (13) | 5 (12)

12. Primary Outcome: Change in Visual Acuity From Baseline to 1 Year Grouped by Diffuse vs. Focal Edema as Characterized by the Investigator
Description: as for outcome 3
Time Frame: from baseline to 1 Year
Measure: Mean (Standard Deviation); unit: Letters
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
Letters
  Typical/predominantly focal | 3 (13) | 8 (11) | 8 (13) | 3 (11)
  Neither predominantly focal nor diffuse | 2 (14) | 10 (9) | 8 (15) | 3 (13)
  Typical/predominantly diffuse | 3 (13) | 9 (12) | 10 (10) | 5 (14)

13. Secondary Outcome: Number of Laser Treatments Received Prior to the 1 Year Visit
Description: One eye in the sham+prompt laser group did not receive laser until post 1-year due to an adverse event unrelated to study treatment. One eye in the triamcinolone+prompt laser did not receive laser until after 1-year due to missing 2 consecutive visits at the time of required laser treatment.
Time Frame: 1 Year
Population: Number who completed the 1-year visit.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 274 | 171 | 178 | 176
Number analyzed (Eyes) | 274 | 171 | 178 | 176
Eyes
  0 | 1 | 0 | 124 | 1
  1 | 35 | 53 | 36 | 46
  2 | 75 | 54 | 17 | 53
  3 | 107 | 46 | 1 | 49
  4 | 56 | 18 | 0 | 27

14. Other Pre Specified Outcome: Eyes With Alternative Treatments Prior to the 1-year Visit
Description: Each combination of treatment only counted once.
Time Frame: 1 Year
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
Eyes
  Intravitreal bevacizumab | 3 | 0 | 0 | 1
  Intravitreal triamcinolone acetonide | 5 | 0 | 0 | 0
  Vitrectomy | 2 | 0 | 0 | 0
  Intravitreal bevacizumab+triamcinolone acetonide | 4 | 0 | 0 | 0
  Total number of eyes with alternative treatments | 14 | 1 | 0 | 1
  Total number of treatments applied | 25 | 1 | 0 | 1
  Total per protocol treatments applied | 5 | 1 | 0 | 1
  Total deviations from protocol treatments applied | 9 | 0 | 0 | 0

15. Other Pre Specified Outcome: Change From Moderately Severe Non-proliferative Diabetic Retinopathy or Better From Baseline to 1-year
Description: 113 eyes had missing or ungradable photos at 1 year. Criteria are based on the ETDRS fundus photographic risk factors for the progression of diabetic retinopathy. ETDRS report no. 12. Ophthalmology 1991; 98:823-833
Time Frame: from baseline to 1 Year
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham | Ranibizumab | Triamcinolone
Number analyzed (Participants) | 150 | 182 | 80
Number analyzed (Eyes) | 150 | 182 | 80
Eyes
  Improved by 2 or more levels | 6 | 46 | 20
  Worsened by 2 or more levels | 11 | 5 | 2
Statistical Analysis 1: Comparison: Sham vs Ranibizumab; P value for comparison with sham; Test type: Superiority or Other; p = 0.08, GEE repeated measures
Statistical Analysis 2: Comparison: Sham vs Triamcinolone; P value for comparison with sham; Test type: Superiority or Other; p = 0.17, GEE repeated measures

16. Other Pre Specified Outcome: Change From Severe Non-proliferative Diabetic Retinopathy or Worse From Baseline to 1-year
Description: Criteria are based on the ETDRS fundus photographic risk factors for the progression of diabetic retinopathy. ETDRS report no. 12. Ophthalmology 1991; 98:823-833, ETDRS Severity Scale = Diabetic retinopathy absent, minimal non-proliferative diabetic retinopathy (PDR), mild to moderately severe non-PDR, severe non-PDR, scars of full pr partial panretinal photocoagulation present PDR absent, mild to moderate PDR, high risk PDR, cannot grade, missing.
Time Frame: from baseline to 1 Year
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham | Ranibizumab | Triamcinolone
Number analyzed (Participants) | 83 | 121 | 70
Number analyzed (Eyes) | 83 | 121 | 70
Eyes
  Improved by 2 or more levels | 10 | 18 | 6
  Worsened by 2 or more levels | 7 | 1 | 2
Statistical Analysis 1: Comparison: Sham vs Ranibizumab; P value for comparison with sham; Test type: Superiority or Other; p = 0.03, GEE repeated measures
Statistical Analysis 2: Comparison: Sham vs Triamcinolone; P value for comparison with sham; Test type: Superiority or Other; p = 0.17, GEE repeated measures

17. Secondary Outcome: Percentage of Eyes Receiving Laser at the 48 Week Visit (%)
Time Frame: 1 Year
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 274 | 171 | 178 | 176
Number analyzed (Eyes) | 274 | 171 | 178 | 176
Eyes | 26 | 16 | 8 | 21

18. Other Pre Specified Outcome: Cardiovascular Events According to Antiplatelet Trialists' Collaboration Through 1 Year
Description: Antiplatelet Trialists' Collaboration is a collaborative overview of randomised trials of antiplatelet therapy - I: Prevention of death, myocardial infarction, and stroke by prolonged antiplatelet therapy in various categories of patients. Antiplatelet Trialists' Collaboration. MBJ 1994; 308:81-106. Nonfatal cerebrovascular accident includes ischemic or hemorrhagic or unknown events. Vascular death includes death from any potential vascular or unknown cause.
Time Frame: 1 Year
Population: Study participants with 2 study eyes are assigned to the non-sham group. Multiple events within a study participant are only counted once per event.
Measure: Number; unit: Participants
Arm/Group | Sham | Ranibizumab | Triamcinolone
Number analyzed (Participants) | 130 | 375 | 186
Participants
  Nonfatal myocardial infarction | 3 | 1 | 2
  Nonfatal cerebrovascular accident | 5 | 3 | 1
  Vascular death | 4 | 7 | 2
  Any ATC cardiovascular event | 10 | 11 | 5

19. Secondary Outcome: Mean Optical Coherence Tomography Retinal Volume at 1 Year
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
mm^3 | 8.1 (1.4) | 7.3 (1.0) | 7.4 (1.2) | 7.5 (1.3)

20. Secondary Outcome: Mean Change in Optical Coherence Tomography Retinal Volume From Baseline to 1 Year
Time Frame: from baseline to 1 Year
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
mm^3 | -1.0 (1.4) | -1.4 (1.4) | -1.5 (1.5) | -1.4 (1.6)
Statistical Analysis 1: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Prompt Laser; Difference in mean change from sham+prompt laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Confidence intervals are adjusted for multiple comparisons; Adjusted for baseline optical coherence tomography (OCT) retinal volume, OCT retinal thickness and visual acuity and correlation between 2 study eyes; Mean Difference (Net) = -0.73, 95% CI 2-sided [-1.01 to -0.44]
Statistical Analysis 2: Comparison: Sham+Prompt Laser vs 0.5 mg Ranibizumab+Deferred Laser; Difference in mean change from sham+prompt laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Confidence intervals adjusted for multiple comparisons; [statistical method as in outcome 20, analysis 1]; Mean Difference (Net) = -0.68, 95% CI 2-sided [-0.96 to -0.41]
Statistical Analysis 3: Comparison: Sham+Prompt Laser vs 4 mg Triamcinolone+Prompt Laser; Difference in mean change from sham+prompt laser; Test type: Superiority or Other; p < 0.001, ANCOVA — Confidence intervals are adjusted for multiple comparisons; [statistical method as in outcome 20, analysis 1]; Mean Difference (Net) = -0.62, 95% CI 2-sided [-0.91 to -0.34]

21. Other Pre Specified Outcome: Major Ocular Adverse Events During First Year of Follow-Up
Time Frame: 1 Year
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sham+Prompt Laser | 0.5 mg Ranibizumab+Prompt Laser | 0.5 mg Ranibizumab+Deferred Laser | 4 mg Triamcinolone+Prompt Laser
Number analyzed (Participants) | 293 | 187 | 188 | 186
Number analyzed (Eyes) | 293 | 187 | 188 | 186
Eyes
  Endophthalmitis | 1 | 1 | 1 | 0
  Pseudoendophthalmitis | 1 | 0 | 0 | 1
  Ocular vascular event | 1 | 1 | 0 | 2
  Retinal detachment | 0 | 0 | 1 | 0
  Vitrectomy | 7 | 0 | 3 | 0
  Vitreous hemorrhage | 15 | 3 | 4 | 2
  Increase in intraocular pressure >=10 mmHg | 16 | 10 | 5 | 70
  Intraocular pressure >=30 mmHg | 3 | 2 | 4 | 46
  Initiation of intraocular lowering medication | 23 | 12 | 7 | 79
  Glaucoma surgery | 0 | 0 | 0 | 0
  Cataract surgery | 11 | 6 | 8 | 19

ADVERSE EVENTS:
Time Frame: 1 Year
Description: All ocular adverse events are listed under treatment group drug. Participants with a systemic adverse event with two study eyes are listed under the sham/ranibizumab or triamcinolone combination.
Groups:
- Sham + Prompt Laser: Laser was given within 3 to 10 days after sham injections, Laser = Focal/grid photocoagulation
- Ranibizumab + Prompt Laser: 0.5 mg intravitreal ranibizumab plus prompt (within 3-10 days after injection) focal/grid photocoagulation
- Ranibizumab + Deferred Laser: 0.5 mg intravitreal ranibizumab with deferred (24 weeks) focal/grid photocoagulation
- Triamcinolone + Prompt Laser: 4 mg intravitreal triamcinolone plus prompt (within 3-10 days after injection) focal/grid photocoagulation
- Sham + Ranibizumab + Laser; Sham + Ranibizumab + Deferred Laser; Sham + Triamcinolone + Laser: Participants in this group had 2 study eyes, the right eye was assigned randomly with equal probability to one of the four groups (Sham + prompt laser, ranibizumab + prompt laser, ranibizumab + deferred laser, triamcinolone + prompt laser). If the right eye was assigned to a treatment group other than the sham + prompt laser group, then the left eye was assigned to the sham + prompt laser group. If the right eye was assigned to the sham prompt + prompt laser group, then the left eye was assigned randomly to one of the other three groups.
Arm/Group | Sham + Prompt Laser | Ranibizumab + Prompt Laser | Ranibizumab + Deferred Laser | Triamcinolone + Prompt Laser | Sham + Ranibizumab + Laser | Sham + Ranibizumab + Deferred Laser | Sham + Triamcinolone + Laser
Serious Adverse Events (participants affected / at risk) | 53/130 | 46/131 | 41/132 | 57/135 | 21/56 | 20/56 | 12/51
Other Adverse Events (participants affected / at risk) | 139/139 | 97/97 | 105/105 | 145/145 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham + Prompt Laser (N=130) | Ranibizumab + Prompt Laser (N=131) | Ranibizumab + Deferred Laser (N=132) | Triamcinolone + Prompt Laser (N=135) | Sham + Ranibizumab + Laser (N=56) | Sham + Ranibizumab + Deferred Laser (N=56) | Sham + Triamcinolone + Laser (N=51)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anemia (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Angina pectoris (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arterial bypass operation (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Vascular disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Blood potassium increased (General disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0
Breast cancer (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 8 | 0 | 4 | 4 | 3 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cellulitis (General disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 0
cerebrovascular accident (Vascular disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 5 | 0 | 3 | 2 | 2 | 0 | 0
Convulsion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Coronary artery disease (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Death (General disorders) | 2 | 1 | 2 | 2 | 1 | 1 | 0
Dehydration (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus inadequate control (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diabetic ketoacidosis (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Dysarthria (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart rate irregular (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (General disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 3 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ischaemic stroke (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leg amputation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 2 | 3 | 2 | 0 | 0
Multiple fractures (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infacrtion (Cardiac disorders) | 3 | 0 | 1 | 2 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural complications (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Presyncope (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 3 | 1 | 1 | 0 | 2 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Shoulder operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Stent placement (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Syncope (General disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endophthalmitis (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Intraocular pressure increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Anxiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biopsy thyroid gland (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Boneneoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric bypass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemiparesis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung cancer metastatic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary gland disorder (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iris neovascularisation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
hypoglycaemia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Anaemia of Chronic disease (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Joint Injury (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin Ulcer (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham + Prompt Laser (N=139) | Ranibizumab + Prompt Laser (N=97) | Ranibizumab + Deferred Laser (N=105) | Triamcinolone + Prompt Laser (N=145) | Sham + Ranibizumab + Laser (N=0) | Sham + Ranibizumab + Deferred Laser (N=0) | Sham + Triamcinolone + Laser (N=0)
Cataract (Eye disorders) | 12 | 9 | 10 | 31 | 0 | 0 | 0
Cataract subcapsular (Eye disorders) | 7 | 5 | 4 | 23 | 0 | 0 | 0
Eye pain (Eye disorders) | 22 | 23 | 20 | 12 | 0 | 0 | 0
Myodesopsia (Eye disorders) | 8 | 4 | 10 | 19 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 9 | 13 | 11 | 23 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 4 | 21 | 25 | 17 | 0 | 0 | 0
Eye Irritation (Eye disorders) | 9 | 8 | 11 | 10 | 0 | 0 | 0
Influenza (General disorders) | 10 | 6 | 6 | 11 | 0 | 0 | 0
Intraocular pressure increased (Eye disorders) | 7 | 4 | 7 | 55 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 9 | 6 | 16 | 5 | 0 | 0 | 0
Maculopathy (Eye disorders) | 24 | 12 | 14 | 9 | 0 | 0 | 0
Nasopharyngitis (General disorders) | 10 | 10 | 10 | 14 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 6 | 10 | 5 | 4 | 0 | 0 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 7 | 6 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 39 | 16 | 20 | 32 | 0 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 13 | 6 | 8 | 11 | 0 | 0 | 0
Visual Disturbance (Eye disorders) | 13 | 7 | 5 | 13 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 15 | 3 | 4 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No